CLINICAL TRIAL: NCT06262061
Title: Propranolol for the Treatment of Traumatic Brain Injury
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Ian Ball, Associate Professor, Department of Medicine, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO-TBI-FS
Record Dates: First submitted 2023-09-21; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: Beta-blockers; TBI; Trauma
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries | interventions — Propranolol

STUDY DESIGN:
Intervention Model Description: Prospective, single- center double- blinded randomized control trial comparing placebo to propranolol for the treatment of moderate- severe traumatic brain injury.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized in a 1:1 allocation to either the propranolol or control group. Our hospital pharmacy will control the randomization procedure. The propranolol group will receive over-encapsulated whole marketed tablets comprised of 20mg oral propranolol [USP grade] filled with lactose monohydrate powder [NF grade] encapsulated with opaque gelatin capsules twice daily for 14 days (or until hospital discharge or death). The control group will receive an oral placebo comprised of lactose monohydrate powder [NF grade] encapsulated with indistinguishable opaque gelatin capsules. The pharmacy will have access to the randomization key. Nursing staff will remove the gelatin capsule casing and dissolve the trial drug & placebo in sterile water prior to administering it enterally via a feeding tube to the participants. Aside from the nursing staff, the participants, research team, and remainder of the clinical care teams will all remain blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol Group (Active Comparator): The propranolol group will receive 20mg of oral propranolol twice daily for 14 days (or until hospital discharge or death).
  Interventions: Drug: Propranolol
- Control Group (Placebo Comparator): Control group will receive an oral placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — 20mg oral propranolol BID x 14 days
  Arms: Propranolol Group
Drug: Placebo — Placebo pill orally BID x 14 days
  Arms: Control Group

SUMMARY:
Traumatic brain injury (TBI) is a leading cause of global disease and directly affects over 1.5 million Canadians, with 165 000 TBIs occurring yearly in Canada. Despite the burden of TBIs, there are limited treatment options available and current treatments generally focus on supportive care. The aim of TBI treatment is reduce inflammation and damage occurring after the TBI (secondary injury).

Beta- blockers (BBs) are medications commonly used to block the actions of endogenous catecholamines- hormones that are thought to contribute to secondary injury within brain tissue. This reduces metabolic demand in the vulnerable, injured brain. BBs have been studied in several retrospective trials and one single-center, non- blinded randomized controlled study. These results point towards a benefit to the use of BBs in TBI but need to be confirmed in a rigorous manner before they are widely adopted.

The current study aims to assess the feasibility of a single centre randomized controlled trial of BBs versus placebo to treat moderate to severe TBI. This feasibility trial will inform the planning of a large multi-center study powered to detect a difference in cognitive outcomes and mortality. It also will allow the investigators to gather biologic samples for measuring serum catecholamines and inflammatory mediators to better understand the basic science mechanisms of BBs in this patient population; and to assess the feasibility of using the Cambridge Battery to assess cognitive outcomes of trial participants.

DETAILED DESCRIPTION:
Traumatic brain injury is a spectrum of illness ranging from mild concussive symptoms to debilitating and even life-threatening injury. Between 2002 and 2016, there were 3550 deaths per year due to TBI. Between 2006 and 2018 there were 17 500 hospitalizations per year due to TBI. As TBIs often affect youth and working- age adults they are responsible for a very large economic burden, costing Canada $7.3 billion in 2011 and rising to a projected $8.2 billion in 2031.

TBI causes morbidity and morbidity in two phases. The primary (initial) injury results in damage to brain tissue, and is only preventable with injury prevention programs. The cornerstone of medical TBI management hinges on avoidance of secondary injury to vulnerable brain tissue. This translates to supportive care for these patients, such as normalization of vital signs, blood glucose and treatment of seizures, if present. Any abnormalities such as low blood pressure or oxygen levels do not provide an appropriate environment for the recovery of brain function and negatively impact recovery. There are few targeted medications that can be given in the initial management of TBI patients. One of these groups of medications is osmotic agents that help to reduce intracranial pressure in cases of elevated intracranial pressure. Osmotic agents, such as mannitol or hypertonic saline, act transiently and as a bridging therapy to surgical intervention. Medications to reduce bleeding, such as TXA, have been studied but have not been shown to reduce mortality. Given the limitations and equivocal role of these medications, additional therapies to reduce the devastating sequelae in TBI patients are necessary.

Beta-blockers are a class of medications which act on various b adrenergic receptors in the body, either b1 or b2. b1 receptors are located primarily in the heart and to a lesser extent the kidneys and adipose tissue; while b2 receptors are located in the lungs, vasculature and liver. Depending on which b receptors are inhibited, different beta-blockers exert variable physiologic effects. There are non-selective beta-blockers (bind to both b1 and b2) as well as selective beta-blockers (solely bind to b1 receptors) available. Propranolol is an example of a non-selective beta-blocker - it will lower heart rate and blood pressure by its cardiac effects on b1 receptors but also acts peripherally. Propranolol can uniquely cross the blood-brain barrier and is able to bind to b receptors that are also present in the central nervous system. TBI patients commonly develop episodes of elevated heart rate, blood pressure and agitation secondary to overactivation of the sympathetic nervous system. Administration of beta-blockers helps mitigate these events, thereby reducing the metabolic demand in vulnerable, injured brain. It is because of these mechanisms that propranolol is the beta-blocker that has been postulated to be most beneficial for patients with TBI. Blocking these receptors leads to decreased metabolic demand and inflammation in neuronal cells. An important objective of this feasibility trial is for the investigator team to collaborate with Dr. Allan and her team to measure differences in serum catecholamines and inflammatory mediators between participants in the Propranolol group as compared to the placebo group.

There have been several retrospective analyses of patients with TBI on at-home beta-blocker therapy or who received beta-blockers during the course of their hospital stay, many of which demonstrated improved outcomes. In a meta-analysis combining prospective and retrospective cohorts, beta- blocker administration was associated with a reduction in in-hospital mortality. The only randomized control study of propranolol in TBI examined early administration of propranolol to TBI patients and its impacts on plasma catecholamine levels and physiologic parameters. The authors found lower levels of plasma catecholamines and improved vital signs, including Glasgow Coma Scale (GCS) scores at 7 days. This study was unblinded and occurred in a single, center and as such is at risk of bias.

While most studies of propranolol in TBI have focused on mortality as the outcome of choice, this is not ideal for several reasons. Mortality is a crude marker of function in TBI, whereas functional outcomes are the patient-centered outcome of choice in neurologic injury. The Glasgow Outcomes Scale (Extended) is a validated measure of neurologic function and is the standard for assessment of recovery following neurological injury.

Additionally, the investigators propose to evaluate the feasibility of using the Cambridge Battery developed by Dr. Adrian Owen to evaluate short and longer term cognitive outcomes in trial participants. This neuropsychologic measure has been used in a variety of neurologic testing studies evaluating CNS disorders and medication, but has not to date been applied to TBI patients. This represents an exciting opportunity to develop a new tool for the assessment of the traumatically brain injured patient, with the advantage of a strong record of safety and reliability in other populations.

In order to change practice, an adequately powered, multi-center RCT is necessary to evaluate the role of beta-blockers in patients with TBI. The investigators propose a feasibility study of beta-blockers in TBI at London Health Sciences Center (LHSC) as a first step towards a future multi-center RCT.

ELIGIBILITY:
Inclusion Criteria

1. Adult patients (>18/= 18 years of age) who have sustained a TBI
2. Initial GCS during the first 6 hours of assessment of 5- 12 (inclusive)

Exclusion Criteria

1. Home beta- blocker therapy
2. New indication for beta- blocker therapy during hospital stay
3. Contraindication to beta- blocker therapy

   1. Allergy
   2. Severe asthma/ COPD
   3. Sinus bradycardia and greater than first degree block
   4. Patients in cardiogenic shock
   5. Right ventricular failure secondary to pulmonary hypertension
   6. Congestive heart failure unless the failure is secondary to a tachyarrhythmia treatable with propranolol
4. Patients requiring any vasoactive medications to maintain their blood pressure at the time of enrollment
5. Patients requiring or are on any of the following medications:

   1. Digitalis
   2. Anesthetic agents that maintain cardiac contractility by virtue of their effect on catecholamine release (e.g., ether)
   3. Epinephrine, noradrenaline, adrenaline, and isoproterenol
   4. Antiarrhythmic cardiac depressant drugs such as procainamide or quinidine
   5. Thiazide-like diuretics and/or peripheral vasodilators
   6. Catecholamine depletion drugs such as reserpine or guanethidine
6. Patients not expected to survive 48 hours
7. >24 hours from trauma at the time of enrollment

   a. Patients on vasoactive medications at initial trial screening may enter the trial if their vasopressor requirements cease within 24 hours of their trauma
8. Inability to secure enteral access for medication administration
9. Doses of BB will be held under the following circumstances

   a. HR <45 or MAP <55 for 5 minutes prior to administration time
10. Patients that are pregnant and/or breastfeeding participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Hospital Mortality | 1 month
Cognitive function | 6 months
  Assessment of neurological function at time of discharge, 2 week follow-up, and 6 month follow-up using Glascow Outcome Scale Extended (GOS-E) and Cambridge Battery via a validated online platform

SECONDARY OUTCOMES:
Catecholamines/Inflammatory markers | patient's blood will be drawn to measure the 5 serum biomarkers on admission and then at 24hr, 48hrs, 72 hours and 5 days following the initial TBI injury
  We will measure five TBI serum markers (S100B, NSE, GFAP, UCH-L1 and TAU).

IPD SHARING:
Plan to Share IPD: No